CLINICAL TRIAL: NCT01825044
Title: An Open-label, Uncontrolled Phase II-study to Investigate Pharmacokinetics, Safety and Biomarkers of Effectiveness of NeuroSTAT® (Ciclosporin) in Patients With Severe Traumatic Brain Injury (TBI)
Brief Title: Copenhagen Head Injury Ciclosporin (CHIC) Study
Acronym: CHIC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NeuroVive Pharmaceutical AB (Industry)
Responsible Party: Sponsor
Organization: Abliva AB (Industry)
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2012.001; 2012-000756-34 (EudraCT Number)
Record Dates: First submitted 2013-03-20; First posted 2013-04-05 (Estimated); Last update posted 2017-10-04 (Actual); Status verified 2017-10

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic Brain Injury; TBI; ciclosporin; pharmacokinetic; safety; microdialysis; mitochondrial protection
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NeuroSTAT 5 mg/kg/day (Active Comparator): Intravenous bolus of NeuroSTAT (Ciclosporin) 2.5 mg/kg bodyweight followed by 5 days of 5 mg/kg bodyweight/day continuous infusion
  Interventions: Drug: NeuroSTAT 5 mg/kg/day
- NeuroSTAT 10 mg/kg/day (Active Comparator): Intravenous bolus of NeuroSTAT (Ciclosporin) 2.5 mg/kg bodyweight followed by 5 days of 10 mg/kg bodyweight/day continuous infusion
  Interventions: Drug: NeuroSTAT 10 mg/kg/day

INTERVENTIONS:
Drug: NeuroSTAT 5 mg/kg/day — Intravenous bolus of NeuroSTAT (Ciclosporin) 2.5 mg/kg bodyweight followed by 5 days of 5 mg/kg bodyweight/day continuous infusion
  Other Names: Ciclosporin 5 mg/kg/day
  Arms: NeuroSTAT 5 mg/kg/day
Drug: NeuroSTAT 10 mg/kg/day — Intravenous bolus of NeuroSTAT (Ciclosporin) 2.5 mg/kg bodyweight followed by 5 days of 10 mg/kg bodyweight/day continuous infusion
  Other Names: Ciclosporin 10 mg/kg/day
  Arms: NeuroSTAT 10 mg/kg/day

SUMMARY:
This is an open label study on the pharmacokinetics and safety of ciclosporin in patients with severe traumatic brain injury, who require intensive care unit admission and monitoring of intracranial pressure via a ventricular catheter. 20 patients will be screened, and subsequently enrolled after clinical stabilisation. Thereafter, patients will receive 2.5 mg/kg bolus dose infusion of ciclosporin, followed by either 5 mg/kg/day or 10 mg/kg/day of ciclosporin as continuous infusion for 5 days+3 days monitoring at the intensive care unit. After an additional 30 days, a follow-up phone call will be made to the patient, or the patient's nursing staff, checking patient status and serious adverse events. The two dose levels will be investigated in 10 patients each, starting with the lower dose level for the first 10 patients. Patients will have samples of blood and cerebrospinal fluid drawn at pre-defined time points during the study for pharmacokinetic assessment and evaluation of biomarkers. Bedside monitoring with microdialysis and brain tissue oxygenation will be performed. The safety monitoring includes nephrotoxicity, hepatotoxicity, monitoring of intracranial pressure (ICP), infections monitoring and adverse events collection and reporting.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients, age between 18 and 75 years, inclusive.
2. Requirement for Intensive Care Unit (ICU) admission and clinical indication for External Ventricular Drainage (EVD) and Intracranial Pressure (ICP) monitoring.
3. Evidence of non-penetrating severe TBI, confirmed by history and abnormalities consistent with a non-penetrating trauma on computerised tomography (CT) scan upon admission.
4. Clinical examination with post-resuscitation Glasgow Coma Scale (GCS) of 4-8, inclusive.
5. Hemodynamically stable after resuscitation (systolic blood pressure (SBP) >100 mm Hg).
6. Informed consent for participation waived: obtained by two independent physicians and subsequently, the patient's Legally Acceptable Representative (LAR) and General Practitioner (GP). If GP is unavailable, the Danish Health and Medicines Authority can give consent together with the LAR.

Exclusion Criteria:

1. Bilaterally fixed dilated pupils.
2. Penetrating traumatic brain injury.
3. Spinal cord injury.
4. Pure epidural haematoma.
5. Currently developed, known or a medical history of renal disorder, significant renal failure, or high risk renal failure, defined as:

   1. Serum creatinine ≥ 1.5 x upper limit of normal (ULN).
   2. Pre-existing chronic renal failure with estimated glomerular filtration rate (eGFR)< 60 ml/min/1.73m2 estimated by the simplified Modification of Diet in Renal Disease (MDRD) Study formula.
   3. Major rhabdomyolysis with serum creatine kinase > 5,000 IU/L.
   4. Renal injury resulting in loss of a kidney (either due to direct trauma or ischaemia).
   5. Vascular injury with renal ischaemia likely to cause an episode of acute renal failure.
   6. Any history of renal replacement therapy.
6. Known or a medical history of hepatic disease.
7. Prolonged and/or uncorrectable hypoxia, as judged by the investigator (PaO< 60 mmHg) or hypotension (SBP< 90 mmHg) upon admission.
8. Suspected or confirmed pregnancy (positive urine sample,followed by confirmational serum human chorionic gonadotropin (HCG) pregnancy test).
9. Immunosuppression due to drugs (for ex. ciclosporin) or disease (e.g. human immunodeficiency virus (HIV), malignancy).
10. Known or a medical history of serious chronic viral or fungal infection.
11. Known or a medical history of active mycobacterial infection or antituberculous treatment.
12. Known or a medical history of any allergic reactions and/or anaphylactic reactions towards ciclosporin, egg, peanuts or soya-bean proteins.
13. Ongoing preinjury therapy with any of these drugs:

    rosuvastatin, tacrolimus, Hypericum perforatum (St.John´s Wort; a herbal dietary supplement), stiripentol, aliskiren, bosentan, diltiazem, verapamil and antiepileptics.
14. Participation in other clinical trials.
15. Any significant disease or disorder including abnormal laboratory tests which, in the opinion of the investigator, may either put the patient at risk because of participation in the study, or may influence the results of the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2017-09-21 (Actual); Study Completion 2017-09-21 (Actual)

PRIMARY OUTCOMES:
Non-compartmental analysis of pharmacokinetics (PK) of Ciclosporin in whole blood | Prespecified timepoints during 8 days (PK)
  Peak Plasma Concentration (Cmax) of Ciclosporin and Area under the blood concentration versus time curve (AUC) of Ciclosporin. This will characterise the pharmacokinetic profile of the two chosen dosing regimens of ciclosporin in severe Traumatic Brain Injury (TBI) patients.
Incidence of adverse events | 38 days
  Including:
  1. Ciclosporin levels in whole blood.
  2. Markers of nephrotoxicity: plasma creatinine plasma Cystatin-C and blood urea nitrogen.
  3. Markers of hepatotoxicity: prothrombin time (PT), aspartate transaminase (AST), alanine transaminase (ALT) and bilirubin.
  4. Intracranial Pressure (ICP)
  5. Assessment of infections: according to standard procedures at intensive care unit.

SECONDARY OUTCOMES:
Ciclosporin levels in cerebrospinal fluid (CSF) | Prespecified timepoints during 8 days
  The CSF samples will be drawn from the EVD-catheter at the same time points as in blood to document central nervous system penetration of ciclosporin
Safety biomarkers for nephrotoxicity | Measured at prespecified timepoints during 8 days
  Kidney Injury Molecule (KIM)-1, creatinine and Cystatin-C in urine samples

OTHER OUTCOMES:
Electroencephalography (EEG). | During 8 days
  The background pattern will be interpreted and analysed by an EEG program. The aim is to find evidence if EEG analyses could be used to predict clinical outcome.
Biomarkers of brain injury in brain tissue | Measured at prespecified timepoints during 8 days
  Microdialysis in the most and least traumatised side pre-treatment and every second hour until the end of day 8
Brain tissue oxygen | During 8 days
  Continuously (every 5th second) measured directly using an indwelling probe.

CONTACTS AND LOCATIONS:
Overall Officials: Jesper Kelsen, MD., PhD, Principal Investigator — Dept. of Neurosurgery, Rigshospitalet, Copenhagen, Denmark
Locations (1):
- Dept. of Neurosurgery, Rigshospitalet, University of Copenhagen, Copenhagen, Denmark

REFERENCES:
- [Derived] Hansson MJ, Elmer E. Cyclosporine as Therapy for Traumatic Brain Injury. Neurotherapeutics. 2023 Oct;20(6):1482-1495. doi: 10.1007/s13311-023-01414-z. Epub 2023 Aug 10. PMID 37561274